CLINICAL TRIAL: NCT00180245
Title: Tumor Metabolism of Head and Neck Cancer in Patients Who Underwent Radiation Therapy Measured With F-18-FDG-PET
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Jörg Kotzerke, Prof. Dr., Technische Universität Dresden
Other Study IDs: HNO-FDG-FU
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Cancer
Keywords: Radiation therapy; F-18-FDG
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to describe the regional and global FDG-kinetics in head and neck cancer during percutaneous radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed head and neck cancer not curable by surgery
* Karnofsky > 70%
* Tumor volume and localization allow curative radiotherapy
* Written consent

Exclusion Criteria:

* Metastases
* Earlier radiotherapy of head or neck
* Pregnancy
* Secondary malignancy excluding dermal carcinoma T1 and Tis-carcinoma of cervix uteri
* Psychiatric impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes consecutive patients from the Department of Radiooncology with head and neck cancer (HNC) intended for a curative chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2005-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Kotzerke, MD, Principal Investigator — Department of Nuclear Medicine
Locations (1):
- Department of Nuclear Medicine, Dresden, Germany